CLINICAL TRIAL: NCT04845321
Title: Phase 1 Study to Evaluate the Safety and Pharmacokinetics of Single and Multiple Ascending Doses of VNRX-9945 in Healthy Adult Volunteers
Brief Title: VNRX-9945 Safety and Pharmacokinetics in Healthy Adult Volunteers
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Part 2 terminated, unrelated to safety.
Sponsor: Venatorx Pharmaceuticals, Inc. (Industry)
Collaborators: Novotech (Australia) Pty Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Basic Science
Other Study IDs: VNRX-9945-101
Record Dates: First submitted 2021-04-10; First posted 2021-04-14 (Actual); Last update posted 2025-06-10 (Actual); Status verified 2025-06

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VNRX-9945 (Experimental): Oral dosing
  Interventions: Drug: VNRX-9945
- Placebo (Placebo Comparator): Oral dosing
  Interventions: Drug: Placebo for VNRX-9945

INTERVENTIONS:
Drug: VNRX-9945 — Part 1: One dose except food effect cohort (receives two doses) Part 2: 14 doses (once a day for 14 days)
  Arms: VNRX-9945
Drug: Placebo for VNRX-9945 — Part 1: One dose except food effect cohort (receives two doses) Part 2: 14 doses (once a day for 14 days)
  Arms: Placebo

SUMMARY:
This is a 2-part first-in-human dose-ranging study to evaluate the safety and pharmacokinetics of escalating doses of VNRX-9945.

DETAILED DESCRIPTION:
In Part 1, subjects will receive a single dose of VNRX-9945 or placebo. Subjects enrolled in the food effect cohort will receive a dose in a fasted and fed state (total 2 doses) of VNRX-9945 or placebo following an appropriate washout period between the doses. In Part 2, subjects will receive doses of VNRX-9945 or placebo daily for 14 days.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults 18-55 years
2. Males or non-pregnant, non-lactating females
3. Body mass index (BMI) between 18 and 32.0 kg/m2 and total body weight >50 kg (110 lbs)
4. Normal blood pressure
5. Normal lab tests

Exclusion Criteria:

1. Current cardiovascular, respiratory, hepatic, renal, gastrointestinal, endocrine, autoimmune, hematologic, neoplastic, or neurological disorder
2. History of severe allergic or anaphylactic reaction
3. Abnormal ECG or history of clinically significant abnormal rhythm disorder
4. Positive alcohol, drug, or tobacco use/test

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2021-06-23 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
Part 1: Number of subjects with adverse events | Up to 8 days after last administration of study drug
Part 2: Number of subjects with adverse events | Up to 8 days after last administration of study drug

SECONDARY OUTCOMES:
Part 1: AUC0-tau | Days 1-6 (Days 1-12 for fasted/fed cohort)
Part 1: Cmax | Days 1-6 (Days 1-12 for fasted/fed cohort)
Part 1: tmax | Days 1-6 (Days 1-12 for fasted/fed cohort)
Part 1: AUCinf | Days 1-6 (Days 1-12 for fasted/fed cohort)
Part 1: t1/2 | Days 1-6 (Days 1-12 for fasted/fed cohort)
Part 2: AUC0-tau | Day 1 and Following Last Dose on Day 14
Part 2: Cmax | Day 1 and Following Last Dose on Day 14
Part 2: tmax | Day 1 and Following Last Dose on Day 14
Part 2: t1/2 | Following Last Dose on Day 14

CONTACTS AND LOCATIONS:
Locations (1):
- New Zealand Clinical Research, Auckland, New Zealand